CLINICAL TRIAL: NCT07085637
Title: Intravenous Hydrogen Nanobubbles Effect on Cardiac Physiology and Quality of Life: a Single Blind, Dose-response Study
Brief Title: IV Hydrogen Nanobubbles for Cardiac Function and QoL
Acronym: HNB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia Molecule Institute (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: No. 410/KPEK-POLKESMA/2022
Record Dates: First submitted 2025-06-02; First posted 2025-07-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases; Hypertension; Blood Pressure
Keywords: hydrogen nanobubbles; cardiovascular physiology; health-related quality of life; blood pressure; myocardial relaxation
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of the following six groups, with interventions administered intravenously twice a week over a 5-week period. Group A is the control group; intervention of intravenous 500 mL of normal saline (NS) for 10 sessions over 5 weeks. Group B; intervention of 5 mL of HNB in NS i.v. for 10 sessions over 5 weeks. Group C with 10 mL HNB, group D 15 mL, group E 20mL, and group F with 25mL HNB, all done in 10 sessions over 5 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Different dosage types (Experimental): This study was designed as a randomized, single-blind, dose-response clinical trial consisting of six distinct arms. The first arm served as the control group, where participants received 500 mL of normal saline without any hydrogen nanobubbles, functioning as a placebo. The remaining five arms were intervention groups that received intravenous infusions of hydrogen nanobubbles (HNBs) at different doses. Specifically, participants in Arm B received 5 mL of HNB, Arm C received 10 mL of HNB, Arm D received 15 mL of HNB, Arm E received 20 mL of HNB, and Arm F received 25 mL of HNB, with each dose diluted in normal saline.
  All participants underwent a total of 10 infusion sessions over a period of 5 weeks, receiving treatments twice weekly. The study was conducted under single-blind conditions. This multi-arm design allowed the researchers to systematically evaluate the dose-dependent effects of HNB therapy on cardiovascular function, blood biomarkers, and health-related quality of life.
  Interventions: Other: intravenous infusion of hydrogen nanobubbles (HNB) administered twice weekly over a 5-week period

INTERVENTIONS:
Other: intravenous infusion of hydrogen nanobubbles (HNB) administered twice weekly over a 5-week period — This study investigated a novel intervention using intravenous hydrogen nanobubbles (HNBs), which are microscopic hydrogen gas bubbles encapsulated in liquid, offering enhanced stability, deep tissue penetration, and sustained antioxidant and anti-inflammatory effects. Unlike other hydrogen therapies (such as inhalation or hydrogen-rich water), this method delivers HNBs directly into the bloodstream.
  Participants were randomized into six groups: one control group receiving saline and five intervention groups receiving escalating doses of HNBs (5-25 mL) over 10 intravenous infusions in 5 weeks. This intervention is distinct for its dose-response design, intravenous delivery, and combined evaluation of cardiovascular function and quality of life (SF-36)-a patient-centered approach not commonly found in similar studies.

SUMMARY:
The goal of this clinical trial is to learn if intravenous hydrogen nanobubbles (HNBs) improve cardiovascular function and quality of life in adults. It will also explore the dose-dependent effects of HNBs when given through IV infusion.

The main questions it aims to answer are:

1. Do HNBs improve heart function and blood vessel health (e.g., blood pressure, ejection fraction, flow-mediated dilation)?
2. How do different doses of HNBs affect quality of life as measured by the SF-36 questionnaire?
3. Are there any safety or tolerability concerns with intravenous HNBs?

Researchers will compare different doses of HNBs (5 mL to 25 mL) to a placebo (normal saline) to evaluate their physiological and psychological effects. Participants will:

1. Receive intravenous infusions twice a week for 5 weeks (10 sessions in total)
2. Be assigned randomly to one of six groups (five different HNB doses or placebo)
3. Complete quality-of-life questionnaires and undergo cardiovascular and lab tests before and after the intervention

DETAILED DESCRIPTION:
This clinical study explored whether intravenous hydrogen nanobubbles (HNBs) can improve heart health and quality of life. HNBs are microscopic hydrogen gas bubbles that may help reduce oxidative stress and inflammation-two major contributors to cardiovascular disease. The research aimed to assess how different doses of HNBs affect blood pressure, heart function, blood vessel health, and overall well-being.

A total of 52 healthy adults aged 18-65 took part in the trial. They were randomly assigned to receive either normal saline (as a placebo) or saline mixed with varying doses of HNBs (5-25 mL). Each participant received 10 intravenous infusions over 5 weeks, with health checks before and after. Researchers used physical exams, blood tests, heart scans, and a standardized questionnaire (SF-36) to track changes in cardiovascular function and quality of life.

This study helps lay the groundwork for future research into non-drug therapies using nanotechnology. If proven effective, HNBs could become a novel, low-risk treatment option for people with high blood pressure, heart stress, or chronic inflammation-ultimately supporting both physical and emotional well-being.

ELIGIBILITY:
Inclusion Criteria

Participants will be eligible for inclusion in the study if they meet all of the following criteria:

1. Aged between 18 and 65 years at the time of screening.
2. Demonstrated stable health condition, as determined by medical history and baseline clinical evaluation.
3. Willing and able to provide written informed consent.
4. Able to comply with study procedures and agree to maintain normal daily activities and dietary patterns throughout the study period.

Exclusion Criteria

Participants will be excluded from the study if they meet any of the following criteria:

1. Known or suspected hypersensitivity to hydrogen or hydrogen-based products.
2. Current participation in another interventional clinical trial.
3. Diagnosed with advanced or uncontrolled cardiovascular, renal, or hepatic disease.
4. Any other medical or psychological condition that, in the opinion of the investigators, could compromise the participant's safety or the integrity of the study data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Physiology | From enrollment to the end of treatment at 6 weeks
  Primary cardiovascular function outcomes included systolic and diastolic blood pressure, measured in millimeters of mercury (mmHg); heart rate, expressed in beats per minute (bpm); and left ventricular ejection fraction (LVEF), reported as a percentage. Diastolic function was assessed through early diastolic mitral inflow velocity (EVel), lateral mitral annular velocity (ELat), and septal mitral annular velocity (ESep), all expressed in meters per second (m/s). Left Ventricular Mass divided by Body Surface Area (BSA) to report Left Ventricular Mass Index in (g/m²), relative wall thickness (RWT), presented as a unitless ratio; tricuspid annular plane systolic excursion (TAPSE), interventricular septal thickness in diastole (IVSd), left ventricular internal dimension in diastole (LVIDd), and left ventricular posterior wall thickness in diastole (LVPWD), all reported in centimeters (cm).Flow-mediated dilation (FMD) (% change in vessel diameter)
Health-Related Quality of Life (HRQoL) | From enrollment to the end of treatment at 6 weeks
  The study evaluated health-related quality of life (HRQoL) using the 36-Item Short Form Health Survey (SF-36), a validated instrument consisting of eight distinct domains: General Health (GH), Physical Functioning (PF), Role Limitations due to Physical Health (PH), Bodily Pain (BP), Vitality (VT), Social Functioning (SF), Role Limitations due to Emotional Problems (EL), and Mental Health (MH). Each domain was treated as a separate outcome measure and scored individually on a scale from 0 to 100, where higher scores reflect better health status in that specific domain. In accordance with reporting standards, each SF-36 domain was analyzed and reported independently, rather than being combined into a single summary score. Although all domains share the same unit (0-100 scale), they assess different dimensions of physical and mental well-being and are therefore presented as distinct outcome variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Indonesia Molecule Institute, Malang, East Java, Indonesia

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT07085637/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT07085637/ICF_001.pdf